CLINICAL TRIAL: NCT01612364
Title: Double-Blind Randomized Controlled Trial: Thoracic Sympathetic Block for the Treatment of Complex Regional Pain Syndrome I of the Upper Limb
Brief Title: RCT :Thoracic Sympathetic Block for the Treatment of Complex Regional Pain Syndrome I of the Upper Limb
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Roberto O Rocha, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5138 - 1805142/1
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Complex Regional Pain Syndrome I of Upper Limb
Keywords: CRPS I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thoracic sympathetic block (Experimental): Sympathetic block of upper limb via thoracic vertebra T3
  Interventions: Procedure: thoracic sympathetic block
- control block (Active Comparator): Same medication used in experimental group, but in dorsal subcutaneous
  Interventions: Procedure: thoracic sympathetic block

INTERVENTIONS:
Procedure: thoracic sympathetic block — Thoracic sympathetic block is sympathetic block of upper limb described by Leriche e Fontaine em 1925. The block is performed under radioscopic view, positioning the needle lateral the body of thoracic vertebra T3, where infuse anesthetic solution. The theoretical advantage over the stellate ganglion is its greater specificity and efficiency. Solution block: 5ml ropivacaine 0,75% + 5ml de triamcinolone 2%
  Other Names: T2-T3 thoracic sympathetic block; T3 sympathetic block; T2-T3 thoracic dorsal sympathetic block; thoracic sympathetic ganglion block

SUMMARY:
This is a double-blind randomized controlled trial to evaluate the efficacy of the sympathetic block via thoracic vertebra T3 for the treatment of CRPS I upper limb. Patients with CRPS I refractory to medical treatment will be subjected to four physical therapy sessions and then the randomized for experimental or control block and then more four physiotherapy sessions. Patients will be evaluated after one month of the blockade (primary outcome) and then up to 12 months. Will be evaluated by analgesic scale (Mcgill, brief pain inventory, dn4 questionnaire, NPSI, VAS), functional (ADM) and quality of life (HAD and WHOQOL-brief).

ELIGIBILITY:
Inclusion Criteria:

* Complex regional pain syndrome (IASP, 1994) involving an upper limb;
* Pain scores in excess of five visual analog scale (VAS);
* Poor outcome to treatment (less than 50% reduction in VAS scores) -

Exclusion Criteria:

* History of severe brain injury, epilepsy and stroke
* Patients who had undergone sympathetic ganglion block for treatment of the affected limb, by any technique
* Severe systemic disease
* Addictive behavior, severe psychiatric disorders, psychiatric diseases untreated
* Refusal to participate or not initial adherence to orientations
* Refusal to be randomized in a treatment group or with contraindications to any of them pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Analgesia after block | 1 month
  Analgesia (Mcgill, brief pain inventary, DN4 questionaire, VAS) and functional (ADM) evaluation.

SECONDARY OUTCOMES:
analgesia quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roberto O Rocha, MD, Principal Investigator — Hospital das Clinicas Faculty of Medicine University Sao Paulo
Locations (1):
- Hospital das Clinicas, Faculty of Medicine, University of Sao Paulo, São Paulo, São Paulo, Brazil